CLINICAL TRIAL: NCT05904886
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Study Evaluating Atezolizumab and Bevacizumab, With or Without Tiragolumab, in Patients With Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: A Study Evaluating Atezolizumab and Bevacizumab, With or Without Tiragolumab, in Participants With Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma (HCC) (IMbrave152)
Acronym: SKYSCRAPER-14
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CO44668; 2023-503422-39-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-05-23; First posted 2023-06-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Tiragolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study has been unblinded as of amendment version 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Bevacizumab + Tiragolumab (Experimental): Atezolizumab plus bevacizumab plus tiragolumab will be administered every 3 weeks (Q3W) until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Tiragolumab
- Atezolizumab + Bevacizumab + Placebo (Placebo Comparator): Atezolizumab, bevacizumab plus placebo will be administered Q3W until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Other: Placebo

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 milligrams (mg) on Day 1 of each 21-day cycle.
  Other Names: Tecentriq; MPDL3280A; RO5541267
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a dose of 15 milligrams per kilogram (mg/kg) on Day 1 of each 21-day cycle.
  Other Names: Avastin
Drug: Tiragolumab — Tiragolumab will be administered by IV infusion at a fixed dose of 600 mg on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A; RO7092284
  Arms: Atezolizumab + Bevacizumab + Tiragolumab
Other: Placebo — Placebo matching tiragolumab will be administered by IV infusion on Day 1 of each 21-day cycle.
  Arms: Atezolizumab + Bevacizumab + Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of tiragolumab, an anti-TIGIT monoclonal antibody, when administered in combination with atezolizumab and bevacizumab as first-line treatment, in participants with unresectable, locally advanced or metastatic HCC.

Per amendment version 5, following a memo issued by the Sponsor, participants receiving treatment in the atezolizumab plus bevacizumab plus tiragolumab arm are recommended to discontinue tiragolumab treatment unless the investigator decides the benefit outweighs the risk. Participants receiving treatment in atezolizumab plus bevacizumab plus placebo arm must discontinue placebo treatment. Participants may continue receiving active treatment(s) per protocol until loss of clinical benefit or unacceptable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology/cytology or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic participants
* Disease that is not amenable to curative surgical and/or locoregional therapies
* No prior systemic treatment for locally advanced or metastatic and/or unresectable HCC-measurable disease according to RECIST v1.1
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1 within 7 days prior to randomization
* Child-pugh Class A within 7 days prior to randomization
* Adequate hematologic and end-organ function
* Female participants of childbearing potential must be willing to avoid pregnancy within 5 months after the final dose of atezolizumab, within 6 months after the final dose of bevacizumab, and within 90 days after the final dose of tiragolumab/placebo
* Male participants with a female partner of childbearing potential or pregnant female partner must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of bevacizumab and for 90 days after the final dose of tiragolumab/placebo to avoid exposing the embryo.

Exclusion Criteria:

* Pregnancy or breastfeeding within 5 months after the final dose of atezolizumab, within 6 months after the final dose of bevacizumab, and within 90 days after the final dose of tiragolumab/placebo
* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with locoregional therapy to liver within 28 days prior to initiation of study treatment, or non-recovery from side effects of any such procedure
* Treatment with systemic immunostimulatory agents
* Treatment with systemic immunosuppressive medication
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Mixed histology or other subtypes/variants of HCC, including, but not limited to, known liver adenocarcinoma, fibrolamellar HCC, sarcomatoid HCC, other rare HCC variant, or mixed cholangiocarcinoma and HCC
* Co-infection with hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Acute epstein-barr virus (EBV) infection or known or suspected chronic active EBV infection
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From randomization to the first occurrence of disease progression (PD) or death from any cause, whichever occurs first (up to approximately 21 months)
Overall Survival (OS) | From randomization to death from any cause (up to approximately 36 months)

SECONDARY OUTCOMES:
Investigator-assessed Confirmed Objective Response Rate (ORR) According to RECIST v1.1 | From randomization up to approximately 21 months
Investigator-assessed Duration of Response (DOR) According to RECIST v1.1 | From the first occurrence of a documented confirmed objective response to the first occurrence of PD or death from any cause, whichever occurs first (up to approximately 21 months)
Investigator-assessed PFS Rate According to RECIST v1.1 at 6 and 12 Months | Month 6, Month 12
OS Rate at 1 and 2 Years | Year 1, Year 2
Investigator-assessed PFS According to HCC mRECIST | From randomization to the first occurrence of PD or death from any cause, whichever occurs first (up to approximately 21 months)
Investigator-assessed Confirmed ORR According to HCC mRECIST | From randomization up to approximately 21 months
Investigator-assessed DOR According to HCC mRECIST | From the first occurrence of a documented confirmed objective response to the first occurrence of PD or death from any cause, whichever occurs first (up to approximately 21 months)
Time to Confirmed Deterioration (TTCD) Assessed Using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer 30 (EORTC QLQ-C30) Subscales | Up to approximately 21 months
  The following subscales of the EORTC QLQ-C30 will be used for the assessment: global health status/quality-of-life (GHS/QoL), physical functioning and role functioning. GHS and QoL are scored on a 7-point scale: 1=Very poor to 7=Excellent. Functioning items are scored on a 4-point scale: 1=Not at all to 4=Very much, with a higher score indicating a worse outcome. Scores will be linearly transformed with a minimum score of 0 and maximum score of 100. A higher score indicates a better outcome.
Change from Baseline in GHS/QoL, Physical Functioning, and Role Functioning Assessed Using the EORTC QLQ-C30 | Up to approximately 21 months
  GHS and QoL are scored on a 7-point scale: 1=Very poor to 7=Excellent. Functioning items are scored on a 4-point scale: 1=Not at all to 4=Very much, with a higher score indicating a worse outcome. Scores will be linearly transformed with a minimum score of 0 and maximum score of 100. A higher score indicates a better outcome.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 36 months
Serum Concentrations of Atezolizumab | Prior to the first infusion and 30 minutes after atezolizumab infusion on Day 1 of Cycle 1 (cycle = 21 days), prior to infusion on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit (up to approximately 21 months)
Serum Concentrations of Tiragolumab | Prior to the first infusion and 30 minutes after tiragolumab infusion on Day 1 of Cycle 1 (cycle = 21 days), prior to infusion on Day 1 of Cycles 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit (up to approximately 21 months)
Percentage of Participants With Anti-drug Antibodies (ADAs) to Tiragolumab | Prior to the first infusion on Day 1 of Cycles (cycle = 21 days) 1, 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit (up to approximately 21 months)
Percentage of Participants With ADAs to Atezolizumab | Prior to the first infusion on Day 1 of Cycles (cycle = 21 days) 1, 2, 3, 4, 8, 12, 16 and at treatment discontinuation visit (up to approximately 21 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (171):
- United States (34):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - UCSF Fresno at Community Cancer Institute, Clovis, California
  - City of Hope Cancer Center, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Va Palo Alto Health Care System, Palo Alto, California
  - UCLA Cancer Center, Santa Monica, California
  - Hartford Healthcare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - University of Illinois, Chicago, Illinois
  - Norton Cancer Institute - Audubon, Louisville, Kentucky
  - Ochsner Cancer Inst., New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Minnesota Oncology Hematology Woodbury, Woodbury, Minnesota
  - Washington Uni School of Medicine, St Louis, Missouri
  - NYU Langone, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - James J Peters VA Hospital / Mental Illness Research Education and Clinic Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Thomas Jefferson Uni, Philadelphia, Pennsylvania
  - North Texas VA Medical Center, Dallas, Texas
  - Kelsey Seybold Clnic, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Inst., Seattle, Washington
  - Univ of Wisconsin-Madison, Madison, Wisconsin
- Belgium (3):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (8):
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Oncoclínicas do Brasil - BELO HORIZONTE, Belo Horizonte, Minas Gerais
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro
- Canada (4):
  - Juravinski Hospital, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- China (22):
  - Baoji Central Hospital, Baoji
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Peoples Hospital of Hunan Province, Changsha
  - Hunan Cancer Hospital, Changsha
  - West China Hospital - Sichuan University, Chengdu
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Provincial People?s Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Lishui Central Hospital, Lishui
  - Zhongshan Hospital Fudan Unvierstiy, Shanghai
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Xi'an Inernational Medical Center Hospital, Xi'an
- Côte d’Ivoire (2):
  - Polyclinique Internationale Sainte Anne- Marie (PISAM), Abidjan
  - Centre National d'Oncologie Médicale et de Radiothérapie Alassane Ouattara (CNRAO), Abidjan
- France (10):
  - CHU CAEN - Hôpital de la Côte de Nacre, Caen
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hopital Dupuytren, Limoges
  - Fondation Hopital Saint Joseph, Marseille
  - Hopital Hotel Dieu Et Hme, Nantes
  - APHP - Hopital Saint Antoine, Paris
  - Hopital Robert Debre, Reims
  - Centre Hospitalier Valence, Valence
  - Hopitaux de Brabois - Gastro-Entereologie, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
- Germany (4):
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinikum Magdeburg Klinik für Gastroenterologie und Hepatologie, Magdeburg
  - Uniklinik Mainz, Mainz
  - Universität Tübingen, Tübingen
- Ghana (2):
  - KBTH, Accra
  - Sweden Ghana Medical Center, Accra
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hosp, Shatin
- Italy (7):
  - Az. Osp. G. Panico, Tricase, Apulia
  - A.O. S. Orsola Malpighi, Bologna, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Az. Osp. Uni Ria San Martino, Genoa, Liguria
  - IRCCS Istituto Clinico Humanitas, Rozzano, Lombardy
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - A.O.U.I. Verona-Ospedale Policlinico G.B. Rossi Borgo Roma, Verona, Veneto
- Japan (20):
  - Fujita Health University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital East, Chiba
  - Ehime Prefectural Central Hospital, Ehime
  - Kurume University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Sapporo Kosei General Hospital, Hokkaido
  - Hokkaido University Hospital, Hokkaido
  - Kanazawa University Hospital, Ishikawa
  - Toranomon Branch Hospital, Kanagawa
  - Kanagawa Cancer Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Iwate Medical University Hospital, Numakunai
  - The University of Osaka Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Jichi Medical University Hospital, Tochigi
  - Toranomon Hospital, Tokyo
  - Japanese Red Cross Musashino Hospital, Tokyo
- University of Nairobi - Institute of Tropical and Infectious Diseases, Nairobi, Kenya
- Mexico (4):
  - OncoMed, Mexico City, Mexico CITY (federal District)
  - Centro Medico Nacional Siglo Xxi - Imss, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Ciencias Médicas Y de Nutricion Salvador Zubirán, Mexico City, Mexico CITY (federal District)
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington
- Nigeria (2):
  - Jos University Teaching Hospital, Jos
  - Lagos University Teaching Hospital Lagos (LUTH), Lagos State, Lagos
- Poland (2):
  - ID Clinic, Mysłowice
  - NIO im Marii Sklodowskiej-Curie, Warsaw
- PanOncology Trials, San Juan, Puerto Rico
- National Cancer Centre, Singapore, Singapore
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Limpopo Cancer Research Institute, Polokwane
- South Korea (8):
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (11):
  - Hospital de Navarra, Navarra, Navarre
  - Clinica Universitaria de Navarra, Pamplona/iruña, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universitaria de Navarra de Madrid;Servicio de Hepatologia, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Clinico de Valencia, Valencia
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Centre, Tainan
  - National Taiwan Uni Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Khon Kaen Uni, Khon Kaen
- Turkey (Türkiye) (5):
  - Adana Baskent University Medical Faculty, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Gazi Uni Medical Faculty Hospital, Ankara
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - ?zmir Medical Point, Kar?iyaka
- Uganda Cancer Institute, Kampala, Uganda
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - Royal Free Hospital, London
  - Hammersmith Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Badhrinarayanan S, Cotter C, Zhu H, Lin YC, Kudo M, Li D. IMbrave152/SKYSCRAPER-14: a Phase III study of atezolizumab, bevacizumab and tiragolumab in advanced hepatocellular carcinoma. Future Oncol. 2024;20(28):2049-2057. doi: 10.1080/14796694.2024.2355863. Epub 2024 Jun 10. PMID 38861301